CLINICAL TRIAL: NCT04865510
Title: Citrate Versus Heparin in Continuous Renal Replacement Therapy : Effect on Cardiovascular System and Clot Circuit in Critically Ill Patients
Brief Title: Citrate Versus Heparin in Continuous Renal Replacement Therapy :
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Collaborators: King Chulalongkorn Memorial Hospital (Other); Chiang Mai University (Other); Department of Medicine, Somdech Phra Pinklao Hospital, Bangkok, Thailand. (Unknown)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: COA033/61
Record Dates: First submitted 2021-04-22; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Acute Kidney Injury; Citrate; Cytokines; Hemodynamic Responses
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: This study is a prospective,multicenter, open-label randomized trial
Who Masked: Care Provider
Masking Description: systemic random sampling (block of four). Group A was the citrate group while group B was heparin- free method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Citrate (Active Comparator): The RCA group CRRT were performed with Prisma flex or (Baxter Healthcare/Gambro Spain) or Informed machine with citrate pump. The function mode was continuous venovenous hemodiafiltration (CVVHDF) in postdilution mode with ST 150 filter sets. The substitution fluid was Accusol or Prismocal B22 .The dose of dialysis was 20-25 ml/kg/hr with blood flow 150-200 ml/min. Trisodium citrate solution (4%,136mmol/L) was infused into the arterial line prior to the blood pump at a dose of 4 mmol/L of plasma flow. Calcium chloride (5% 340 mmol/L elemental calcium) was infused into the venous return to maintain systemic ionized calcium in the normal range (0.99-1.30 mmol/L) and the targets values for ionized calcium (iCa2+) after the dialysis membrane were 0.25-0.35 mmol/L. The rale of calcium infusion was adjusted in a timely manner based on repeated measurements of calcium concentration
  Interventions: Procedure: Regional citrate anticoagulation
- Heparin-free (Placebo Comparator): The heparin- free group The circuit was periodically flushed with 50 ml saline via access limb every 30 minutes .When pre-filter pressure started to rise, additional saline flushes would be given.
  Interventions: Procedure: Regional citrate anticoagulation

INTERVENTIONS:
Procedure: Regional citrate anticoagulation — The investigators collected patient's plasma at study start (day 0) and at day 3, 5, 7, 14, 28) .Samples were used to measure inflammatory markers (Il 6, IL 8, IL 10 and TNFα) .
  . Markers of dialysis efficiency (BUN, creatinine) and other parameters related to AKI (acid base status, calcium, phosphorus, hemoglobin). The recorded variables also included adverse events, dialysis clotting, hemodynamic status, duration of mechanical ventilation, inotropic support. The hemodynamic parameters were monitored by EV 1000 clinical platform .The investigators measured cardiac performance data, which includes cardiac output (CO), cardiac index (CI), stroke volume (SV), and stroke volume indexes (SVI). Moreover, it also provides information about systemic vascular resistance (SVR). Thus, patient hemodynamic parameters as mentioned above were measured at the following 6 time-point: after the initiation of CRRT (T1), every 6 hours later for 24 hours (T2, T3, T4, T5), and at hour-72 (T6).
  Other Names: Heparin-free

SUMMARY:
This study is a prospective, multicenter, open-label randomized trial comparing regional citrate anticoagulation (RCA) with heparin-free protocol. The function mode was continuous venovenous hemodiafiltration (CVVHDF) in post-dilution mode. The investigators measured hemodynamic changes at certain time points after starting CRRT (0, 6, 12, 24, 48, 72 hr).Levels of inflammatory cytokine (IL-1β, IL-6, IL-8, IL-10 and TNF-ɑ) were measured at day 1 and day 3

DETAILED DESCRIPTION:
Twenty patients were randomized into heparin group and 11 patients were in citrate group. The cardiac performance were not significantly different between 2 groups at every time point. The inflammatory cytokines declined similarly in both treatment arms. The maximum filter survivial time was longer in a RCA group but not reach statistically significant (44.64±26.56 hr vs p=0.693 in citrate and heparin free group respectively).There was no serious side effects dung both treatment arm even in the group of liver dysfunction patients.

ELIGIBILITY:
Inclusion Criteria:

* need for CRRT,
* no contraindication to CRRT

Exclusion Criteria:

* patients with previous history of chronic kidney disease (CKD) (baseline serum creatinine > 2 mg/dL (male) or > 1.5 mg/dL (female)
* history of renal transplantation
* known pregnancy
* previous dialysis within 30 days
* severe liver disease
* end stage heart disease or untreatable malignancy
* moribund patients with expected survival less than 30 days
* previous use of heparin or other anticoagulant, antiplatelet within 7 day except use for deep vein thrombosis
* active bleeding at the time of enrollment and/or severe coagulopathy
* receiving blood or blood components prior to enrollment
* hemoglobin less than 7.5 g/dL and/or platelet count less than 100,000/mm3
* previous underlying clotting disorders such as hypercoagulable state
* severe malnutrition (Body mass index (BMI ) less than 18)
* underwent CRRT for other reasons besides acute kidney injury (AKI)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Cardiac output | 72 hour
  cm3/min
Cardiac index | 72 hour
  L/min/m2
Systemic vascular resistance | 72 hour
  mmHg⋅min⋅mL-1
Systemic vascular resistance index | 72 hour
  dynes · sec/cm5/m2

SECONDARY OUTCOMES:
Filter life span | through study completion,an aveage of 72 hours
  Hours of filter use
Changes of IL-1β | day 1,day 3
  Unit/ml
Changes of IL-6 | day 1,day 3
  Unit/ml
Changes of IL-8 | day 1,day 3
  Units/ml
Changes of IL-10 | day 1,day 3
  Units/mL
Changes of TNF-ɑ | day 1,day 3
  Uniys/mL
Mortality | 28 day
  patient survival
Renal survival | 28 day
  dialysis dependent

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, M.D., Principal Investigator — Renal unit,Faculty of Medicine,Vajira Hospital,Navamindradhiraj University
Locations (1):
- Faculty of Medicine ,Vajira hospital,Navamindradhiraj University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Oudemans-van Straaten HM, Kellum JA, Bellomo R. Clinical review: anticoagulation for continuous renal replacement therapy--heparin or citrate? Crit Care. 2011 Jan 24;15(1):202. doi: 10.1186/cc9358. PMID 21345279
- [Result] Gatward JJ, Gibbon GJ, Wrathall G, Padkin A. Renal replacement therapy for acute renal failure: a survey of practice in adult intensive care units in the United Kingdom. Anaesthesia. 2008 Sep;63(9):959-66. doi: 10.1111/j.1365-2044.2008.05514.x. Epub 2008 Jun 28. PMID 18549413
- [Result] Borg R, Ugboma D, Walker DM, Partridge R. Evaluating the safety and efficacy of regional citrate compared to systemic heparin as anticoagulation for continuous renal replacement therapy in critically ill patients: A service evaluation following a change in practice. J Intensive Care Soc. 2017 Aug;18(3):184-192. doi: 10.1177/1751143717695835. Epub 2017 Mar 14. PMID 29118829
- [Result] Cutts MW, Thomas AN, Kishen R. Transfusion requirements during continuous veno-venous haemofiltration: -the importance of filter life. Intensive Care Med. 2000 Nov;26(11):1694-7. doi: 10.1007/s001340000676. PMID 11193279
- [Result] Morabito S, Pistolesi V, Tritapepe L, Fiaccadori E. Regional citrate anticoagulation for RRTs in critically ill patients with AKI. Clin J Am Soc Nephrol. 2014 Dec 5;9(12):2173-88. doi: 10.2215/CJN.01280214. Epub 2014 Jul 3. PMID 24993448
- [Result] Tuerdi B, Zuo L, Sun H, Wang K, Wang Z, Li G. Safety and efficacy of regional citrate anticoagulation in continuous blood purification treatment of patients with multiple organ dysfunction syndrome. Braz J Med Biol Res. 2017 Nov 17;51(1):e6378. doi: 10.1590/1414-431X20176378. PMID 29185591
- [Result] Schrezenmeier EV, Barasch J, Budde K, Westhoff T, Schmidt-Ott KM. Biomarkers in acute kidney injury - pathophysiological basis and clinical performance. Acta Physiol (Oxf). 2017 Mar;219(3):554-572. doi: 10.1111/apha.12764. Epub 2016 Aug 25. PMID 27474473
- [Result] Kwon O, Molitoris BA, Pescovitz M, Kelly KJ. Urinary actin, interleukin-6, and interleukin-8 may predict sustained ARF after ischemic injury in renal allografts. Am J Kidney Dis. 2003 May;41(5):1074-87. doi: 10.1016/s0272-6386(03)00206-3. PMID 12722043
- [Result] Liangos O, Kolyada A, Tighiouart H, Perianayagam MC, Wald R, Jaber BL. Interleukin-8 and acute kidney injury following cardiopulmonary bypass: a prospective cohort study. Nephron Clin Pract. 2009;113(3):c148-54. doi: 10.1159/000232595. Epub 2009 Aug 12. PMID 19672112
- [Result] de Fontnouvelle CA, Greenberg JH, Thiessen-Philbrook HR, Zappitelli M, Roth J, Kerr KF, Devarajan P, Shlipak M, Coca S, Parikh CR; TRIBE-AKI Consortium. Interleukin-8 and Tumor Necrosis Factor Predict Acute Kidney Injury After Pediatric Cardiac Surgery. Ann Thorac Surg. 2017 Dec;104(6):2072-2079. doi: 10.1016/j.athoracsur.2017.04.038. Epub 2017 Aug 16. PMID 28821332
- [Derived] Trakarnvanich T, Sirivongrangson P, Trongtrakul K, Srisawat N. The effect of citrate in cardiovascular system and clot circuit in critically ill patients requiring continuous renal replacement therapy. J Artif Organs. 2023 Mar;26(1):53-64. doi: 10.1007/s10047-022-01329-0. Epub 2022 Apr 12. PMID 35412099